CLINICAL TRIAL: NCT05680649
Title: Effect of Breathing Exercise During Peripheral Intravenous Catheter Implementation on Pain, Anxiety, and Patient Satisfaction
Brief Title: Effect of Breathing Exercise During Peripheral Intravenous Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Instructor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 573/2022
Record Dates: First submitted 2022-12-15; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Venipuncture
Keywords: Anxiety; Breathing exercise; Nursing; Pain; peripheral intravenous catheterization
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Breathing exercise
  Interventions: Other: Breathing exercise
- Control (No Intervention): Standard practice

INTERVENTIONS:
Other: Breathing exercise — Diaphragmatic breathing exercises were taught to the individuals by the researcher and they were asked to start breathing exercises before starting PIVC. While the PIVC was being placed, the individuals continued the breathing exercise and the breathing exercise was terminated at the end of the application.
  Arms: Intervention

SUMMARY:
This study was carried out to determine the effect of breathing exercise performed during peripheral intravenous catheter (PIVC) application on pain, anxiety and patient satisfaction.

The study was completed as a randomized controlled experimental study with a total of 130 individuals who met the inclusion criteria. The Descriptive Characteristics Questionnaire, the State-Trait Anxiety Inventory, and the Numerical Rating Scale were used to collect the data of the study. In addition, Algometer (66 Lb/30 Kg) device was used to evaluate the pain pressure threshold in determining the individuals to be included in the research sample. The individuals in the intervention group were given diaphragmatic breathing exercise while applying the catheter, and the individuals in the control group were inserted without any application.

DETAILED DESCRIPTION:
This study was carried out to determine the effect of breathing exercise performed during peripheral intravenous catheter (PIVC) application on pain, anxiety and patient satisfaction.

The study was completed as a randomized controlled experimental study with a total of 130 individuals who met the inclusion criteria, 65 of whom were in the intervention group and 65 in the control group. Ethics committee approval, institutional permission, and written informed consent from individuals were obtained in the study. The Descriptive Characteristics Questionnaire, the State-Trait Anxiety Inventory, and the Numerical Rating Scale were used to collect the data of the study. In addition, Algometer (66 Lb/30 Kg) device was used to evaluate the pain pressure threshold in determining the individuals to be included in the research sample. The individuals in the intervention group were given diaphragmatic breathing exercise while applying the catheter, and the individuals in the control group were inserted without any application.

ELIGIBILITY:
Inclusion Criteria:

* able to speak and understand Turkish,
* between the ages of 18-65,
* having orientation to place and time,
* without any psychiatric disease and hearing problems,
* not using central nervous system drugs,
* people who having PIVC indication,
* no analgesic or anesthetic agent was applied 24 hours before PIVC application,
* not have any pain in any part of the body that may affect the results of the study,
* no PIVC experience in the last month,
* 20-G catheter will be applied,
* pressure pain threshold mean of 8-16 pounds (Lb), (11) individuals who volunteered to participate in the study.

Exclusion Criteria:

* Infection in the area where PIVC will be applied, -having previous operation, scarring, psoriasis, active dermatitis in the area - -
* where PIVC will be applied,
* with peripheral nerve disease,
* no catheter applied to the forearm veins,
* having diabetes,
* with peripheral neuropathy,
* diagnosed with cancer,
* receiving cancer treatment,
* with respiratory disease,
* who have an obstacle to breathing exercise,
* in the post-surgical period,
* individuals who did not volunteer to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Pain level | 3 minutes after catheter insertion
  Pain level measured with Numeric Rating Scale. The number "0" on the scale means that they do not feel any pain and the number "10" refers to the worst pain.
Anxiety level | 3 minutes after catheter insertion
  Anxiety level measured with Numeric Rating Scale. The number "0" on the scale means that they do not feel any anxiety and the number "10" refers to the highest level of anxiety.

SECONDARY OUTCOMES:
Satisfaction level | 3 minutes after catheter insertion
  Satisfaction level measured with Numeric Rating Scale. The number "0" in the scale indicates that the participants are not at all satisfied with the application, and the number "10" indicates the highest level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Korkut, Study Director — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozkan O, Korkut S. Effect of Breathing Exercise During Peripheral Venous Catheterization on Pain, Anxiety, and Patient Satisfaction: A Randomized Controlled Trial. J Perianesth Nurs. 2024 Aug;39(4):630-637. doi: 10.1016/j.jopan.2023.11.006. Epub 2024 Feb 29. PMID 38430076